CLINICAL TRIAL: NCT03243032
Title: Pain Management Using Pre-Emptive Analgesia in Dental Implant Surgery - A Randomized, Double-Blind, Placebo-Controlled, Clinical Trial
Brief Title: Pre-Emptive Analgesia in Dental Implant Surgery
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: IRB requirements to start study could not be met in a timely manner
Sponsor: Satheesh Elangovan (Other)
Responsible Party: Sponsor-Investigator, Satheesh Elangovan, Principal Investigator, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201707814
Record Dates: First submitted 2017-07-26; First posted 2017-08-08 (Actual); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Ibuprofen; Anti-Inflammatory Agents, Non-Steroidal; Anesthesia

STUDY DESIGN:
Intervention Model Description: Randomized, parallel arms, double-blinded, placebo-controlled trial
Who Masked: Participant
Masking Description: Patients will not know which arm they will be in initially. At the 2 week post-operative visit they may be notified of which arm they participated in if they so choose to find out.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Local Anesthetic Group 1 (Experimental): Group 1 (Pre-emptive analgesia with long acting local anesthesia - experimental group): Ibuprofen 600mg given 30 minutes prior to beginning of surgery. Surgery will be performed only using 0.5% bupivacaine with 1:200,000 epinephrine as the local anesthetic. Following the procedure, all patients will be prescribed Chlorhexidine rinse ( 0.12%) (Rinse with 15 ml two times a day and spit) for 10 days and Antibiotics: Amoxicillin 500 mg three times a day for 7 days or if allergic to penicillin, clindamycin 300 mg four times a day for 7 days. Ibuprofen (600 mg) q 6 hours: prn for pain will be provided to all patients at no charge. Tramadol 50 mg (one every 4-6 hours as needed for pain; maximum 400 mg/day) for uncontrolled pain.
  Interventions: Drug: Ibuprofen 600 mg; Drug: Local anesthetic Group 1
- Local Anesthetic Control (Placebo Comparator): Group 2 (Control / standard of care group): Placebo oral capsule (Microcrystalline Cellulose NF (Avicel PH 105) - compounded at the University of Iowa College of Dentistry Pharmacy) given 30 minutes prior to beginning of surgery. Surgery will be performed using 2% lidocaine with 1:100,000 epinephrine as the local anesthesia. Following the procedure, all patients will be prescribed Chlorhexidine rinse ( 0.12%) (Rinse with 15 ml two times a day and spit) for 10 days and Antibiotics: Amoxicillin 500 mg three times a day for 7 days or if allergic to penicillin, clindamycin 300 mg 4 times a day for 7 days. Ibuprofen (600 mg) q 6 hours: prn for pain will be provided to all patients at no charge. Tramadol 50 mg (one every 4-6 hours as needed for pain; maximum 400 mg/day) for uncontrolled pain.
  Interventions: Drug: Placebo oral capsule; Drug: Local anesthetic Control

INTERVENTIONS:
Drug: Ibuprofen 600 mg — Ibuprofen 600mg given 30 minutes prior to beginning of surgery
  Other Names: non-steroidal anti-inflammatory (NSAID)
  Arms: Local Anesthetic Group 1
Drug: Local anesthetic Group 1 — 0.5% bupivacaine with 1:200,000 epinephrine as the local anesthetic for Group 1 Experimental.
  Other Names: anesthesia
  Arms: Local Anesthetic Group 1
Drug: Placebo oral capsule — Placebo (Microcrystalline Cellulose NF (Avicel PH 105) - compounded at the University of Iowa College of Dentistry Pharmacy) given 30 minutes prior to beginning of surgery
  Other Names: Placebo - Microcrystalline Cellulose NF (Avicel PH 105)
  Arms: Local Anesthetic Control
Drug: Local anesthetic Control — 2% lidocaine with 1:100,000 epinephrine as the local anesthetic for Group 2 - Control
  Other Names: anesthesia
  Arms: Local Anesthetic Control

SUMMARY:
To determine the clinical effectiveness of combined use of pre-emptive analgesia and long acting anesthesia for pain suppression following dental implant surgery as measured by a validated numerical rating scale and the information related to consumption of post-operative medications.

DETAILED DESCRIPTION:
Dental practitioners often prescribe opioids for the relief of moderate - severe acute post-operative pain.1 There is evidence that alternative approaches, such as the use of long acting local anesthetics along with the combination of non-opioid analgesics such as acetaminophen and nonsteroidal anti-inflammatory drugs (NSAIDs), may prevent the need for opioid medications. With the current national opioid overdose epidemic, government officials have introduced new prescribing recommendations for the management of acute pain. Dentists can play a role to address this epidemic by wider recognition and adoption of the new prescribing recommendations for fast acting pre-emptive non-opioid analgesics to prevent acute dental pain.2 Dentists are the fifth leading prescribers of opioids among health care professionals accounting for 12% of the total immediate-release opioids prescribed in the United States (U.S).3 With the increasing trends of opioid prescribing for dental surgeries in the past few decades, dental implant procedures hold the highest increasing rate for opioid prescribing.4 In the U.S alone, there has been as many as 183,000 prescription opioid overdose related deaths from 1999 to 2015. Since 1999, the mortality rate from opioid overdose has more than quadrupled.5 With more than 650,000 opioid prescriptions being dispensed daily in the U.S,6 there has been a national call to alter the current prescribing patterns of opioids to ensure appropriate indications and patient selection.7 There are multiple adverse effects that may develop from opioid pain medications: nausea, vomiting, constipation, dizziness, headache.8 However, two major concerns associated with the excessive prescribing of opioids are overdosing leading to life threatening respiratory depression problems and the creation of an environment that fosters the development of opioid dependency, abuse and addiction.8 The U.S. Senate passed the 'Comprehensive Addiction and Recovery Act' of 2016 to combat the opioid epidemic.9 This legislation is designed to prevent opioid-related morbidity and misuse via physician and patient education, risk awareness, proper prescribing practices, and efforts to improve safer handling of prescription opioids.9 NSAIDs are widely used for their anti-inflammatory, pain and fever reducing properties. In the periphery, these drugs interfere with the formation of pro-inflammatory modulating prostaglandins and thromboxane A2 via reversible inhibition of the cyclooxygenase enzymes (Cox-1 and Cox-2). NSAIDs exact their effects through a variety of peripheral and central mechanisms. Their efficacy in the reduction of post-operative pain has been widely documented.10 It has been demonstrated that a single dose of an NSAID (i.e. etoricoxib, ketoprofen, diclofenac potassium, diflunisan, ibuprofen) may provide better acute post-operative analgesia than some commonly prescribed single dose opioids, even when they are prescribed in combination with other NSAIDs.10 There is also sound evidence that some individuals receive synergistic analgesic effects when NSAIDs are combined with acetaminophen.11 However, these effects can vary, as not everyone will achieve adequate pain relief even from the most potent drugs. Simple drug combinations of fast acting anti-inflammatories with acetaminophen can reliably provide successful analgesia for many acute pain patients in reasonably low doses.10 While modern dental literature contains numerous articles that support the tolerability, safety and efficacy of NSAIDs, many dental practices continue to prescribe opioids in cases which would likely respond better to other analgesics. Many dentists still underrate the risks and abuse of opioids. That is why it is important to design and test more lucid protocols for prescribing analgesics in dental care settings.

Severity of post-operative pain in periodontal and dental implant surgery can vary between mild to severe 12,13 and patient-reported outcome measures (PROMs) can be adverse at times.14 There is evidence that straightforward implant placement procedure is a surgical procedure associated with relatively low postoperative pain and pain management following dental implants is usually achieved by the use of drugs such as NSAIDs, acetaminophen, and/or opioids.11,15 Pre-emptive analgesia refers to the reduction of pain severity that occurs post-operatively by suppressing pain pre-emptively prior to the performance of the surgical procedure.16,17 Previous studies have shown the rationale and efficacy of using pre-emptive analgesia in periodontal and oral surgical models.18-25 Long acting local anesthetics such as bupivacaine have been shown to prolong the onset of and suppress postoperative pain better than lidocaine, an intermediate duration anesthetic.26,27 With successful pre-emptive analgesia including NSAIDs and long acting local anesthetics, the need for stronger post-operative analgesics, like opioids, may be significantly decreased.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients 18 years of age and under 65 years of age
* ASA Type I & II
* Single tooth edentulous site requiring dental implant placement without any additional bone or soft tissue augmentation at the time of implant placement
* Patients not requiring use of any form of sedation for dental implant surgery (nitrous, oral or IV sedation)

Exclusion Criteria:

* Hypersensitivity to NSAIDs, salicylates, or microcrystalline cellulose NF (Avicel PH 105)
* Liver disease
* Renal disease
* Hypertension and taking angiotensin-converting-enzyme inhibitors and/or diuretics
* Significant respiratory conditions including acute or severe asthma.
* Cardiovascular disease that will prevent the patient from going through the surgical procedure or consuming the required medications: cardiac disease, cardiomyopathy, cardiac arrhythmias, coronary heart disease, acute MI, angina, history of MI, coronary artery bypass grafting (CABG), Aspirin intake, peripheral vascular disease, cerebral vascular disease (stroke, TIA)
* Gastrointestinal disease including irritable bowel disease and gastric ulcers
* Hematological diseases (coagulopathy, hemophilia or thrombocytopenia)
* Pregnancy/lactation at the time of surgery
* Heavy smoking (>10 cigarettes per day)
* Diabetes
* Allergies or intolerance to ibuprofen, opioids, and local anesthetic (lidocaine and bupivacaine)
* History of recreational drug abuse
* History of heavy alcohol use. Substance Abuse and Mental Health Services Administration (SAMSHA)30 defines heavy alcohol use as binge drinking on 5 or more days in the past month. SAMSHA defines binge drinking as 5 or more alcoholic drinks for males or 4 or more alcoholic drinks for females on the same occasion (i.e., at the same time or within a couple of hours of each other) on at least 1 day in the past month.
* Patients currently taking prescription pain medications or have taken over-the-counter pain medications within 4 days of surgery.
* Patients with drug-drug or drug-disease state interactions
* Other significant medical conditions (not reported above) that are likely to prevent the patient from going through the surgical procedure or consuming the required medications.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2017-10-06 (Actual); Primary Completion 2017-11-06 (Actual); Study Completion 2017-11-06 (Actual)

PRIMARY OUTCOMES:
Post-operative pain as measured by numerical rating scale | 24 hours
  Difference in pain scores between test and control groups during the time points assessed (0 min, 30, 60, 90, 120, 150, 180, 210, 240 minutes and 24 hours) will be analyzed.

SECONDARY OUTCOMES:
Total pain medication consumption between test and control | 14 days
  Difference in pain medication consumption between test and control groups
Time duration to take first pain medication between test and control | 14 days
  Difference in the time duration to take the first post-operative pain medication between test and control groups
Post-operative pain with anterior versus posterior site of surgery | 24 hours
  Within the control and test groups, correlation between sites (anterior versus posterior) and post-operative pain levels
Post-operative pain as it correlates with the duration of the surgical procedure | 24 hours
  The duration of each surgical procedure will be recorded and separate correlation analyses will be performed to assess the correlation between procedural duration and post-operative pain, within each arm of the trial.
Pre-surgical anxiety correlated with post-surgical pain | 24 hours
  Association between pre-surgical anxiety level and post-surgical pain level as measured by the pain scale within the control group, within the test group and together.
Complications following surgery | 14 days
  Any complications encountered from medications

CONTACTS AND LOCATIONS:
Overall Officials: Sathesh Elangovan, BDS, Study Director — University of Iowa College of Dentistry
Locations (1):
- Univerity of Iowa College of Dentsitry Dental Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No